CLINICAL TRIAL: NCT05146713
Title: Effect Of Propolis Nanoparticles Versus Sodium Hypochlorite As Root Canal Irrigant On Postoperative Pain And Bacterial Reduction In Mandibular Premolars With Necrotic Pulps (A Randomized Clinical Trial)
Brief Title: Effect of Propolis Nanoparticles on Postoperative Pain and Bacterial Reduction in Mandibular Premolars
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Mohamed Saleh Elaguizy, Principal Investigator (Endodontic Resident), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3-7-1 CairoU
Record Dates: First submitted 2021-10-17; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis nanoparticles extract solution (Experimental)
  Interventions: Dietary Supplement: Propolis nanoparticles extract solution
- sodium hypochlorite (Active Comparator)
  Interventions: Drug: sodium hypochlorite

INTERVENTIONS:
Dietary Supplement: Propolis nanoparticles extract solution — 20 mg/ml propolis nanoparticles in the form of solution prepared from honeybee from various plants.
  Arms: Propolis nanoparticles extract solution
Drug: sodium hypochlorite — 2.5% sodium hypochlorite (household bleaching agent)
  Arms: sodium hypochlorite

SUMMARY:
The aim of this study is to clinically compare the intensity of post-operative pain and the amount of bacterial reduction after using 20mg/ml propolis nanoparticles extract solution during chemo-mechanical preparation, versus 2.5% NaOCl, in asymptomatic necrotic mandibular premolars treated in a single visit.

ELIGIBILITY:
Inclusion Criteria:

1. Systematically healthy patient (ASA I,II).
2. Age between 20 and 55 years
3. Male or female.
4. Asymptomatic mandibular premolar teeth diagnosed with pulp necrosis with or without apical periodontitis.
5. Radiographic examination using Digora intraoral periapical sensor plate and software (Digora; Soredex, Helsinki, Finland) showing mandibular premolars with (smaller than 3 mm (0-2 mm)) periapical radiolucency.

Exclusion Criteria:

1. Medically compromised patients having significant systemic disorders. (ASA III or IV).
2. History of intolerance to NSAIDS.
3. Teeth with:

   * Immature roots
   * Vital pulp tissues.
   * Association with swelling.
   * Acute peri-apical abscess or acute exacerbation of a chronic abscess.
   * Mobility Grade II or III.
   * Previously accessed or endodontically treated
   * Deep periodontal pockets more than 4 mm
   * Vertical root fractures, coronal perforation, calcification, and external or internal root resorptions.
4. Patients who could not interpret the NRS.
5. Patients with diabetes, immune-compromising, and immunosuppression disease and pregnant women were, also, excluded.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | up to 48 hours postoperatively
  postoperative pain will be marked by the patient using the Numerical rating scale (NRS) chart which is an 11 point scale consisting of numbers from 0 through 10, where: 0: reading represents "no pain" 1-3: readings represent "mild pain" 4-6: readings represent "moderate pain" 7-10: readings represent "severe pain"

SECONDARY OUTCOMES:
Intracanal bacterial load change | Throughout the chemo-mechanical preparation of the canal.
  The intracanal bacterial load change will be determined using agar culture technique by counting the colony forming units per milliliter (CFUs/mL) before and after root canal preparation.
Number of analgesic tablets taken by the patient after endodontic treatment | Up to 48 hours postoperative.